CLINICAL TRIAL: NCT04405921
Title: Hydroxychloroquine, Azithromycin in the Treatment of Covid-19 Pneumonia: A Randomized,Open-label,Controlled Clinical Trial
Brief Title: Hydroxychloroquine, Azithromycin in the Treatment of Covid-19
Acronym: PACTT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hôpital Universitaire Farhat Hached (Other)
Responsible Party: Principal Investigator, Amel Letaief, Professor of infectious diseases, Centre Hôpital Universitaire Farhat Hached
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PACTT
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: SARS-CoV-2 Pneumonia; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine associated to azithromycin (Experimental): Hydroxychloroquine: 200 mg twice a day orally or via gastric tube (total 400 mg/day) for 5 days. Azithromycin: 500 mg at day 1 then 250 mg/day for 4 days. with standard of care in association to treatments.
  Interventions: Drug: Hydroxychloroquine 200 Mg Oral Tablet; Drug: Azithromycin 250 MG
- Hydroxychloroquine with placebo (Active Comparator): Hydroxychloroquine: 200 mg twice a day orally or via gastric tube (total 400 mg/day) for 5 days. with standard of care in association to treatments.
  Interventions: Drug: Hydroxychloroquine 200 Mg Oral Tablet

INTERVENTIONS:
Drug: Hydroxychloroquine 200 Mg Oral Tablet — orally or via gastric tube
  Other Names: Plaquenil
Drug: Azithromycin 250 MG — orally or via gastric tube
  Other Names: Azro 250
  Arms: Hydroxychloroquine associated to azithromycin

SUMMARY:
This study investigates the efficay and tolerance of 5-days course of hydroxychloroquine or hydroxychloroquine and azithromycin of patients with COVID-19 infection. The investigators will undertake a randomized, double-blind, controlled Trial in the region of Sousse Tunisia

DETAILED DESCRIPTION:
There is a critical need to identify effective treatments and a number of molecules have been suggested, but The investigators still do not have enough evidence about their efficacy, to treat COVID-19 pneumonia.

One of the most tested treatments was the use of Chloroquine or Hydroxychloroquine associated or not to azithromycin.

Studies have indicated that chloroquine (CQ) shows antagonism against COVID-19 in vitro. It's known to block virus infection by increasing endosomal pH required for virus/cell fusion, as well as interfering with the glycosylation of cellular receptors of SARS-CoV. It's also demonstrated that CQ functioned at both entry, and at postentry stages of the 2019-nCoV infection in Vero E6 cells. Besides its antiviral activity, CQ has an immune-modulating activity, which may synergistically enhance its antiviral effect in vivo.

However, evidence regarding its effects in patients is limited. Among patients with COVID-19, the use of Hydroxychloroquine (HCQ) could significantly shorten time to clinical recovery (TTCR) and promote the absorption of pneumonia. This result has been presented in a randomized controlled trial using two arms HCQ versus conventional treatment. The beneficial effect of HCQ has been proven among mild severity COVID-19 pneumonia but the sample size of this study was limited to 31 patients in each group.

Gautret et al also reported that HCQ treatment is significantly associated with viral load reduction/disappearance in COVID-19 patients and its effect is reinforced by azithromycin. A study showed that azithromycin concentration in phagocytic cells is 40× to 150× higher than plasma concentrations. However, Gautret study has many limitations including selection biases because of non-randomization, a small sample size, and dropout of six patients from the study.

In terms of treatment duration, there is no study supporting a long course treatment of 10 days versus a short course treatment of 5 days for HCQ. This treatment is known to have a large distribution volume of 73 l/kg and a plasma half life going from 22 days to 123 days. This suggests that a short course treatment of Hydroxychloroquine and/or azithromycin could be as effective as a long course treatment.

On the other hand, there are currently no effective specific antivirals or drug combinations supported by high-level evidence, and The investigators don't know if HCQ could be effective or if it's effectiveness may be improved if it's associated with Azithromycin. In fact, this association can lead to improve pneumonia but can also increase the risk of treatment side effects.

ELIGIBILITY:
Inclusion Criteria:

* PositiveSARS-COV-2 RT-PCR in hospitalized patients in University Hospital Farhat Hached in Sousse Tunisia.
* Had either not received hydroxychloroquine before or had received hydroxychloroquine for at least 1 day and could tolerate a dose of 200 mg of hydroxychloroquine/day.

Exclusion Criteria:

* Unableto take oral medication, pregnancy or breast feeding, immune-compromised patients,
* Contraindicationto the studied medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery at day-14, from the start of treatment. | 14 days
  Clinical recovery is defined as a complete resolution clinical signs appeared during the medical history and related to COVID-19.

SECONDARY OUTCOMES:
Viral Clearance via RT-PCR at day 5- 7-10 and day 14 | 5- 7-10 and day 14
  RT-PCR will be realized in same laboratory

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Farhat Hached, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No